CLINICAL TRIAL: NCT05940090
Title: Correlation of Dermatologist Made Biopsy Decisions With Artificial Intelligence (AI) Assisted Total Body Photography Detection of Outlier Lesions
Brief Title: Correlation of Dermatologist Made Biopsy Decision With AI Assisted Total Body Photography Detection of Outlier Lesions
Status: Completed | Type: Observational
Sponsor: Halcyon Dermatology (Other)
Responsible Party: Sponsor
Other Study IDs: Halc-1-ai
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Skin Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Comparison of outlier analysis with dermatologist made biopsy decisions: Skin lesions recommended for skin biopsy by the dermatologist will be compared to lesions highlighted by the application outlier analysis.
  Interventions: Device: SkinIO

INTERVENTIONS:
Device: SkinIO — The device is simply an application that photographs skin lesions and identifies lesions that may require further examination

SUMMARY:
This research study will determine how a smart phone application (app) for total body photography outlier analysis compares to a dermatologist's decision to biopsy skin lesions.

DETAILED DESCRIPTION:
Informed written consent will be obtained by all study subjects. Each participant will be asked to generate a unique identifier, so their demographic data, medical intake, and study assessments can be stored without any patient identifiers. The unique identifier is the participant's 2-digit day of birth, first 3 initials of their mother's maiden name, and the 4 digits of their birth year. All clinical data will be entered into a de- identified database.

Demographic information including age, gender, ethnicity, collected via medical intake survey at the initial visit. Data from the survey will be associated only with the patient's unique identifiers.

ELIGIBILITY:
Inclusion Criteria:

* Males and females participants in overall good health ages 18 to 85 who have skin lesions

Exclusion Criteria:

* Those who are under 18 or over 85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females participants in overall good health ages 18 to 85 who have skin lesions
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
Dermatologist made biopsy decision compared to AI outlier lesions | Three months
  Patient will undergo total body photography that marks outlier lesions. Without reviewing the photos, a dermatologist will make recommendations for which lesions should undergo skin biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Halcyon Dermatology, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No